CLINICAL TRIAL: NCT02070835
Title: Autologous Skin Cell Versus Classic Skin Grafts in Treatment of Diabetic Foot Ulcers: a Comparative Randomized Controlled Trial
Brief Title: Study of Autologous Skin Cell Treating for Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hu Zhicheng (Other)
Responsible Party: Sponsor-Investigator, Hu Zhicheng, FirstSunYetSen, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYSU-2013-048
Record Dates: First submitted 2014-02-22; First posted 2014-02-25 (Estimated); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic Foot Ulcer; Autologous skin cell
MeSH Terms: conditions — Diabetic Foot | interventions — Skin Transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- autologous skin cell (Experimental): autologous skin cell with skin graft
  Interventions: Device: autologous skin cell
- skin graft (Active Comparator): split-thickness skin graft as control group
  Interventions: Procedure: skin graft

INTERVENTIONS:
Device: autologous skin cell — autologous skin cell and skin graft
  Arms: autologous skin cell
Procedure: skin graft — split-thickness skin graft
  Arms: skin graft

SUMMARY:
Diabetic foot ulcer is one of the refractory wounds and always poses many challenges in clinical practice. This study was conducted to have a prospective, randomised, controlled study compare the safety and efficacy of the autologous skin cell with skin graft (experiment group) with split-thickness skin graft (STSG, control group) alone on treating diabetic foot ulcers.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the effectiveness and safety of autologous skin cell with skin graft (experiment group) vs. skin graft (control group) for the treatment of non-healing diabetic foot ulcers. Our hypothesis is that the methods of experiment group is better than the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years old
* with a diagnosis of type 1 or type 2 diabetes
* who had a diabetic low extremity ulcer last for over 4 weeks
* with a stage 2 by Wagner's scale
* size more than 3 cm2
* absence of vascular reconstruction (ankle brachial indices between 0.7 and 1.2)
* had indications of skin grafting were eligible for inclusion

Exclusion Criteria:

* patients with medical conditions that would impair wound healing (e.g. malignancy, autoimmune disease),
* using corticosteroids or immunosuppressor
* a high anesthesiology or surgical risk
* uncontrolled hyperglycemia (preoperative HbA1c greater than 12.0%)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
healing rate | postsurgery week 4
  the percentage of subjects that achieved complete wound closure by week 4, herein complete wound closure is defined as skin re-epithelialization without drainage or dressing requirements

SECONDARY OUTCOMES:
recurrent rate | postsurgery months 6
  the incidence of ulcer recurrence at months 6. Recurrence will be defined as an ulcer occurring at the same location as the healed study ulcer

OTHER OUTCOMES:
complication rate | postsurgery week 4
  the percentage of subjects that who could not achieved complete wound closure by week 4

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Zhu, PI, Principal Investigator — Department of Burns, The First Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Department of Burn Surgery, The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China